CLINICAL TRIAL: NCT04888923
Title: Natural History of The Human Biological Response to Environmental Exposure and Injury
Status: Recruiting | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000152; 000152-E
Record Dates: First submitted 2021-05-14; First posted 2021-05-17 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01-23

CONDITIONS: Inflammation; Normal Controls; Metabolic Disease
Keywords: Blood Collection; Metabolic Disease; Inflammation; Natural History
MeSH Terms: conditions — Inflammation; Metabolic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Controls: General public population, including females and males, who are over the age of 18, with a mixture of races and ethnicities representative of North Carolina.

SUMMARY:
Background:

Environmental exposures like pollution, diet, and stress can help cause human diseases, or make them worse. Researchers want to better understand how injury and inflammation are caused by these exposures. They want to collect biological and environmental samples and other data. They may use the samples to measure a range of factors, like hormones, toxins, and chemicals. This will help them improve their studies.

Objective:

To identify and understand how environmental exposures contribute to human disease.

Eligibility:

Healthy adults ages 18 and older

Design:

Participants will be screened with questions about their health history, demographics, and medicines they take.

Participants may give blood, hair, stool, saliva, and/or urine samples. They may have a skin punch biopsy to collect skin cells. They may give fingernail or toenail clippings. They may give a sample of exhaled breath.

Participants may give a sputum sample. They will inhale a saline mist and cough mucus into a cup.

Participants may have their nasal passages brushed, scraped, or washed.

Participants may give cheek cell samples. They will swish mouthwash and spit it into a cup.

Participants who produce sperm may give samples.

Participants may have bronchoscopy to collect fluid. A saline solution will be put into their lung and then suctioned out, washing areas of the lung.

Participants may have a pelvic or transvaginal ultrasound. They may have lung function tests.

Participants may collect household dust, urine, or stool at home.

Participants will complete surveys about their health, diet, and exposures.

Participation will last for one or more study visits.

Participants may be contacted in the future to take part in other studies.

DETAILED DESCRIPTION:
Study Description:

Environmental exposures such as pollution, diet, stress, etc. contribute to the development and exacerbation of human disease. Understanding the mechanisms of environmentally induced injury and inflammation will allow us to devise better prophylaxis and treatment measures.

Subjects may undergo sampling of (including but not limited to:) blood, urine, saliva, household dust, cheek cells, hair, nasal cells, stool, nail clippings, exhaled breath condensate, sperm samples, skin cells, and/or sputum etc., and may answer predefined questionnaires regarding health and exposures.

Studies which may be performed on collected material includes establishment of cell cultures and immunologic studies.

Objectives:

Primary Objective: To identify the interaction of host and environmental factors in the response to injury and the development of disease.

Secondary Objectives: To develop better methodological tools in order to quantify host-environmental interactions in health and disease.

Endpoints:

Primary Endpoint: Biological markers of cell/tissue injury and inflammation, such as inflammatory cytokines, intracellular kinases or DNA/RNA damage in association with in vitro or in vivo environmental exposures.

Secondary Endpoints: Diseases or pathological processes (e.g. abnormal laboratory values) associated with environmental exposures.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study.
2. Ability to provide informed consent.
3. Able to read and speak English.
4. Male or female, aged greater than or equal to 18.
5. Able to travel to the NIEHS CRU for study visits.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Not willing to have samples stored for future use.
2. Current pregnancy or lactation, by participant verbal confirmation.
3. Any condition that, in the investigator s opinion, places the participant at undue risk for complications associated with required study procedures.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The general community sample will be from Durham, Raleigh, Chapel Hill and other nearby cities close to the NIEHS Clinical Research Unit (CRU).
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
To identify the interaction of host and environmental factors in the response to injury and the development of disease. | On-going
  To identify the interaction of host and environmental factors in the response to injury and the development of disease.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence S Kirschner, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS Clinical Research Unit (CRU), Research Triangle Park, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Most of the participant data will be utilized by investigators in an aggregate way to validate or invalidate their research.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000152-E.html